CLINICAL TRIAL: NCT06129097
Title: Thyme Honey Mouthwash in Management of Periodontitis in Renal Patients on Hemodialysis: A Randomized Controlled Clinical Trial.
Brief Title: Thyme Honey Mouthwash in Management of Periodontitis in Renal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Asmaa bakr, Lecturer Assistant, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-063
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss; Periodontal Inflammation
Keywords: Thyme honey; Nitric oxide; Hemodialysis; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss; Periodontitis

STUDY DESIGN:
Intervention Model Description: Treatment protocol (for the intervention group):
  * Thyme honey will be applied as oral rinse.
  * Based on this protocol, patients will have oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day.
  * Patients will be instructed to perform thyme honey rinses in the oral mucosa.
  * Patients will be instructed not to swallow the thyme honey oral rinse.
  The control group (placebo):
  Patients in the control arm followed the same protocol with normal saline rinses.
  All patients will receive a course of motivation, oral hygiene instructions (emphasizing proper tooth brushing technique, flossing, interdental brush, and mouthwash usage), scaling, polishing and root debridement with an ultrasonic scaler and Gracey curettes.
Who Masked: Outcomes Assessor
Masking Description: The clinical outcome assessor (A.A) will not be aware of which treatment will be being administered, thus yielding a single-blind controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyme honey mouthwash (Experimental): * Thyme honey will be applied as oral rinse.
  * Based on this protocol, patients will have oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day.
  * Patients will be instructed to perform thyme honey rinses in the oral mucosa.
  * Patients will be instructed not to swallow the thyme honey oral rinse.
  Interventions: Other: Thyme honey mouthwash
- Saline mouthwash (Placebo Comparator): Patients in the control arm followed the same protocol with normal saline rinses.
  Interventions: Other: Thyme honey mouthwash

INTERVENTIONS:
Other: Thyme honey mouthwash — * Thyme honey will be applied as oral rinse.
  * Based on this protocol, patients will have oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day.
  * Patients will be instructed to perform thyme honey rinses in the oral mucosa.
  * Patients will be instructed not to swallow the thyme honey oral rinse.

SUMMARY:
There is a known correlation between oral health and systemic disease. Particularly significant evidences associate periodontal bacteria and tooth loss to systemic disorders and specifically to cardiovascular disease, such as high BP. Furthermore, a correlation between periodontal disease and hypertension has been recently reported ESRD and the medications used by those patients create complications in a variety of systems and organs, which frequently worsens or causes new pathologies in the oral cavity, such as caries, periodontal disease, and different mucosal lesions.

Therefore, the current trial was set up to first evaluate the effect of thyme honey oral rinse in ESRD patients with periodontitis using CAL as a primary objective, and to evaluate the clinical effectiveness of thyme honey oral rinse in ESRD patients with periodontitis on bleeding on probing (BOP) and plaque index, and salivary NO levels as secondary objectives.

DETAILED DESCRIPTION:
Periodontal diseases can be seen in up to 90% of the global population, making it the most common oral disease. In the United States alone, cross-sectional studies show that approximately 50% of adults currently have some form of gingivitis, and up to 80% have experienced some form of periodontal disease in their life. Certain groups have been shown to have an increased incidence of periodontal diseases.

There is a known correlation between oral health and systemic disease . Particularly significant evidences associate periodontal bacteria and tooth loss to systemic disorders and specifically to cardiovascular disease, such as high BP. Furthermore, a correlation between periodontal disease and hypertension has been recently reported.

ESRD and the medications used by those patients create complications in a variety of systems and organs, which frequently worsens or causes new pathologies in the oral cavity, such as caries, periodontal disease, and different mucosal lesions.

The emergence of a chronic systemic inflammatory disease in people with ESRD is a common occurrence. The reasons of this inflammation are most likely multifaceted and complex. A number of illnesses and comorbidities have been identified as potential influencers of an increase in the inflammatory state.

The accelerated periodontal disease with pocket formation, gingival recession, and bone and tooth loss is due not only to inadequate oral hygiene and inflammatory disease burden but also to renal osteodystrophy, high urea concentration, salivary changes in composition and the host factors related to the underlying systemic disease that modify the host response to periodontal infection.

Through nitrate-nitrite reduction, some commensal oral bacteria can supply bioactive NO, essential for the endothelial cell function and regulation of arterial BP.

NO is a free radical and simple gas that is synthesized endogenously by a family of enzymes namely NOSs. Normally, NO is produced from the amino acid L-arginine in the presence of oxygen by eNOS and it has an important role in preserving vascular homeostasis. NO is a multifunctional signaling molecule involved in the maintenance of metabolic and cardiovascular homeostasis and also a potent endogenous vasodilator that suppresses the formation of vascular lesions in atherosclerosis. Imbalance in NO bioavailability is associated with some cardiovascular and metabolic diseases.

Reduction of oxygen provision, such as in the case of myocardial ischaemia, compromises NO synthesis.

Decreased production or activity of NO, due to endothelial dysfunction, is responsible for the pathogenesis of many cardiovascular diseases, including atherosclerosis and CVD such as hypertension, coronary artery disease.

The prospective to restore the oral microbiome by probiotics to increase NO bioavailability represents a new strategy in cardiovascular medicine and dentistry. Therefore, providing NO generation by using nitrite and nitrate may be considered a potential therapeutic approach to the management of resistant hypertensive patients.

The anti-inflammatory properties of thyme extracts due to that thyme exerted a dose-dependent decrease in the production and gene expression of the proinflammatory mediators' tumor necrosis factor (TNF)-α, IL-1B, and IL-6 associated with an increase in the anti-inflammatory IL-10 cytokine secretion in activated macrophages, suggesting beneficial application of thyme honey as an oral health aid.

Thyme honey is an Iranian domestic honey produced from the nectar of different species of thyme plants. Its components are different from thyme extract in quantities. The major constituents of thyme extract are phenolic compounds (such as thymol). However, thyme honey may contain some of these essential oil components at a lower concentration Therefore, the current trial was set up to first evaluate the effect of thyme honey oral rinse in ESRD patients with periodontitis using CAL as a primary objective, and to evaluate the clinical effectiveness of thyme honey oral rinse in ESRD patients with periodontitis on bleeding on probing (BOP) and plaque index, and salivary NO levels as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* - Both genders, aged above 18 years.
* All patients must be clinically diagnosed of ESRD undergoing hemodialysis.
* All patients must have a periodontal disease.
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Patient with history of any serious illness as malignancy, who undergo kidney transplant.
* Patients with any autoimmune disease.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Clinical attachment loss (CAL) | 6 weeks
  With a periodontal probe, PD and CAL will be measured on six locations of the teeth (mesio-buccal/facial, mid-buccal/facial, disto-buccal/facial, mesio-lingual/palatinal, mid-lingual/palatinal, disto-lingual/palatinal).

SECONDARY OUTCOMES:
Bleeding on probing | 6 weeks
  The proportion of bleeding sites 10 second after being stimulated by a standardized manual probe with a controlled force to the bottom of the sulcus/pocket at six locations (mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual, disto-lingual) on all present teeth will be assessed dichotomously as a BOP score on all present teeth
Plaque index | 6 weeks
  presence of plaque is scored on a dichotomous variable and the final score per individual is the sum of the plaque scores divided by the number of surfaces examined.
Salivary Nitric oxide levels | 6 weeks
  • Patients will also be asked to wash their mouths before collecting the samples. Then they will ask to collect the saliva using spitting method in a sterile tube every 1 min for 5 min.

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Ghalwash, Phd, Study Director — The British University in Egypt
Locations (1):
- The British University in Egypt, Cairo, Egypt